CLINICAL TRIAL: NCT05871008
Title: Integrated Actionable Aging Assessment for Cancer Patients Pilot
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 23-0440.cc; P50CA244688 (NIH)
Record Dates: First submitted 2023-04-24; First posted 2023-05-23 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Hodgkin Lymphoma; Kidney Cancer; Leukemia; Lymphoid Leukemia; Multiple Myeloma; Myeloid Leukemia; Monocytic Leukemia; Prostate Cancer; Bladder Cancer
MeSH Terms: conditions — Breast Neoplasms; Hodgkin Disease; Kidney Neoplasms; Leukemia; Leukemia, Lymphoid; Multiple Myeloma; Leukemia, Myeloid; Leukemia, Monocytic, Acute; Prostatic Neoplasms; Urinary Bladder Neoplasms | interventions — Social Determinants of Health

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- IA3-CP with SDoH (Experimental): Assess IA3-CP with SDoH and provide feedback (provider & patient)
  Interventions: Other: Assessment tool IA3-CP with SDoH
- IA3-CP only (Experimental): Assess IA3-CP only without added SDoH and provide feedback (provider & patient)
  Interventions: Other: Assessment tool IA3-CP without SDoH
- Control - usual care (No Intervention): Usual care: Assess IA3-CP without providing the feedback report

INTERVENTIONS:
Other: Assessment tool IA3-CP with SDoH — Each patient randomly assigned to IA3-CP with SDoH study arm will complete a pre-visit assessment tool including SDoH. Feedback is provided to provider and patient.
  Arms: IA3-CP with SDoH
Other: Assessment tool IA3-CP without SDoH — Each patient randomly assigned to IA3-CP only study arm will complete a pre-visit assessment tool excluding SDoH. Feedback is provided to provider and patient.
  Arms: IA3-CP only

SUMMARY:
Aging is the greatest risk factor for cancer incidence and mortality. Geriatric screening is recommended to help with treatment discussions, inform intensity of treatment, and identify supportive care needs. Despite a strong evidence base, geriatric assessments are not implemented routinely in oncologic clinics. Similarly, important information on social determinants of health, mental health, and health behaviors are inconsistently assessed, and almost never in an integrated fashion. In an effort to support clinicians delivering the recommended goal-concordant care, the investigators will integrate assessment of geriatric issues, health behaviors, mental health, and social determinants of health into an efficient, actionable contextual assessment system for older cancer patients called Integrated Aging Assessment for Action for Cancer Patients (IA3-CP). The investigators will use D&I strategies including co-creation engagement approaches and form-function methods to develop workflow processes that feasibly integrate the IA3-CP into usual initial assessment with the oncology team. Our objective is to develop and conduct a randomized pilot of the IA3-CP system and hypothesize that our results will show it can be implemented consistently, acted on, improve quality of care, and enhance patient-provider interactions.

DETAILED DESCRIPTION:
Aging is the greatest risk factor for cancer incidence and mortality. Strong data and expert recommendations support the use of geriatric screening assessments to guide treatment for older adults (>65 years old). Geriatric assessment findings can help in treatment discussions, inform intensity of treatment, and identify supportive care needs. Yet, despite evidenced-based benefits, geriatric assessments are not implemented routinely in oncologic clinics. Similarly, there are strong data and expert recommendations for assessment of social determinants of health (SDoH) and health behaviors, but consistent assessment and action on SDoH and health behaviors is infrequent. Clinicians aiming to deliver recommended goal-concordant care to older patients - which is informed by a patient's frailty, SDoH, health behaviors, and mental health - must act without this important contextual information.

We have identified a pragmatic geriatric screening tool (the G8) and adapted it to a validated patient-reported measure. We aim to integrate the novel, validated, patient reported G8 with the NCI funded, theory driven, evidence-based My Own Health Report (MOHR) system that captures patient reported health behavior, mental health, and social determinants of health (SDoH) through a web-based portal. We will integrate assessment of geriatric issues, health behaviors, mental health, and SDoH into an efficient, actionable contextual assessment system for older cancer patients called Integrated Aging Assessment for Action for Cancer Patients (IA3-CP). We will use D&I strategies including co-creation engagement approaches and form-function methods to develop workflow processes that feasibly integrate the IA3-CP into usual initial assessment with the oncology team. Our objective is to develop and conduct a randomized pilot of the IA3-CP system to determine if it can be implemented consistently, acted on, improve quality of care, and enhance patient-provider interactions.

RATIONALE:

The phrase "you have cancer" lands differently with older patients than it does those younger. The issues of frailty, comorbidity, mental and behavioral health, and SDoH are critical to formulating a personalized cancer treatment approach with an older person as they can't put these conditions "on hold" to focus on a cancer diagnosis. Aging is the greatest risk factor for cancer incidence and mortality, with nearly half of all cancers diagnosed after age 65. There is a clear need to create patient-centered care plans that align care that is medically feasible and aligned with individual patient needs, environment, and preferences.

Geriatric screening and assessment is broadly recommended for the care of older persons with cancer. Similarly, there is strong consensus that SDoH (e.g., food scarcity, medical affordability, safe environments) and health behaviors are key drivers of health disparities. Validated, pragmatic patient-report measures of geriatric issues, health behaviors, and SDoH exist but are seldom consistently assessed in clinical practice, hardly ever in an integrated fashion, and even less seldom acted on. Clinics need efficient, cost-effective tools to screen for and address multiple risks at the same time - technology can provide important efficiencies.

SIGNIFICANCE:

Using age as a primary determinant for cancer treatment puts older adults at risk of under- or over-treatment of cancer. Failure to implement available tools that enhance our ability to tailor care planning to the unique needs of older adults represents a critical gap in patient-centered care.

Implementation of geriatric-specific measures: Oncologists recognize functional assessment as a predictor of future morbidity and mortality risk, so much so that it largely dictates oncology treatment selection, yet are using measures insensitive in an older population. Oncologists will often use clinical gestalt to recommend modified variants of standard treatment. An integrated assessment system can provide actionable, more comprehensive personalized data to the patient and care team.

Geriatric 8: The G8 is a brief geriatric assessment tool that has been broadly validated in the oncology setting to screen for potential frailty and need for a comprehensive assessment. It incorporates functional status, cognition and mental health, and nutritional feedback to form a clinic collected 8-item assessment. To address identified barriers to implementation, the investigators adapted the G8 with input from our Rural Cancer Advisory Board to a patient-reported version. The investigators then pilot tested implementation and validity of the modified G8 in seven clinical environments - primary care and oncology in community and academic settings with excellent results. In parallel, the investigators devised a way to integrate the patient-reported items into the UCHealth EHR for use in clinical care and documentation. The investigators now propose to use similar strategies to integrate the IA3-CP into the EHR.

My Own Health Report (MOHR): MOHR is a patient-centered, web-based health risk assessment and feedback system for unhealthy behaviors, mental health status, and prioritizing patient concerns. MOHR has been used successfully in numerous primary care environments and its use has been found to result in patients feeling more cared for by their clinical team. Our randomized trial found that patients receiving MOHR improved physical activity (p < 0.001) and dietary behaviors (p < 0.001) that increase the risk for many oncology toxicities and significantly increased goal setting during primary care visits. The investigators have recently adapted MOHR to include SDoH such as transportation, food access, medication affordability, safety at home, housing, and financial stability. Much like the geriatric screen, MOHR provides information on health behaviors that may be at risk, especially in an older population more likely to face comorbid conditions.

This proposal will integrate our evidence-based health risk assessment (MOHR) with a geriatric health screener (G8) to assess and address the needs of older adults with cancer. Key challenges to assessment of SDoH and cancer risks are the nonsystematic and separate, non-integrated way these assessments are conducted and the limited time in clinic visits to identify risks, and tailor treatment and goal setting to patient context and priorities. When patients complete our MOHR web-based system, actionable information on health risks and SDoH along with patients' priorities provides for more informed and efficient patient-clinician interactions. This is an example of how well-designed, contextually-appropriate technology developed with patients and clinicians can provide important efficiencies to address clinical and implementation challenges.

In combining the extensive preliminary work in designing the modified G8 and the demonstrated success of the MOHR automated assessment and feedback system with the clinical and methodologic expertise of our team, the investigators are positioned to successfully pilot the IA3-CP in the UCCC. This proposal addresses a clear gap in the needs of older cancer patients and clinical teams and will lead to many future collaborations including a UG3/UH3 MPI pragmatic trial submission.

INNOVATION:

Our proposed feasibility pilot will accelerate the implementation of patient-reported measures to inform care planning for the diverse and at-risk population of older adults with cancer. It will also advance transdisciplinary cancer research by demonstrating integration of multiple risk issues in a pragmatic fashion using innovative D&I science and engagement methods.

ELIGIBILITY:
Inclusion Criteria:

* Age > /= 65
* Patient must agree to participate in all study-related activities
* English or Spanish speaking
* Attending initial visit to oncology

Exclusion criteria

* age < 65
* primary language other than English or Spanish

Ages: 65 Years to 111 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Patient reported receipt of quality illness care | 12 weeks
  Measured by the Patient Assessment of Chronic illness Care (PACIC). The score ranges from 1-5 where higher scores mean a better outcome
Number of referrals made and completed for geriatric, health behavior and SDoH issues | 16 weeks
  Measured by data abstraction from EHR

SECONDARY OUTCOMES:
Discussion of IA3-CP related issues in oncologist-patient encounter | 7 months
  Measured by checklist adapted from the Roter interaction analysis system (RIAS) completed from recorded observation of patient-oncologist meeting
Oncologist utility | 7 months
  Did IA3-CP change your care plan? (yes/no) How helpful was it? (6 pt. scale)
Proportion of patients that use IA3-CP screening tool | 7 months
  Measured by clinic leadership report & observation

CONTACTS AND LOCATIONS:
Overall Officials: Russell E Glasgow, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided